CLINICAL TRIAL: NCT01474473
Title: A Pilot Placebo-Controlled, Randomized and Double Blind Monocenter Study Evaluating CACIPLIQ20 Efficacy On Neuropathic Perforating Foot Ulcer Healing In Diabetic Patients Wearing An Irremovable Windowed Resin Cast
Brief Title: Efficacy Of CACIPLIQ20 On Diabetic Ulcers In Patients Wearing An Nonremovable, Windowed, Fiberglass Cast Boot
Acronym: DIAPLIQ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Organ, Tissue, Regeneration, Repair and Replacement (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CT11Q09UPND
Record Dates: First submitted 2011-10-31; First posted 2011-11-18 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Foot Ulcer; Diabetes Mellitus; Diabetic Neuropathy
Keywords: CACIPLIQ20; Matrix Therapy; Diabetic foot
MeSH Terms: conditions — Foot Ulcer; Diabetes Mellitus; Diabetic Neuropathies; Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CACIPLIQ20 and Cast Boot (Experimental): This arm receives treatment by CACIPLIQ20 application every 3 to 4 days and the wounded leg is held with a nonremovable, windowed, fiberglass Cast Boot.
  Interventions: Device: CACIPLIQ20 and Nonremovable, Windowed, Fiberglass Cast Boot
- Placebo and Cast Boot (Placebo Comparator): This arm receives a placebo (saline solution) every 3 to 4 days and the wounded leg is held with a nonremovable, windowed, fiberglass Cast Boot.
  Interventions: Device: Placebo and Nonremovable, Windowed, Fiberglass Cast Boot

INTERVENTIONS:
Device: CACIPLIQ20 and Nonremovable, Windowed, Fiberglass Cast Boot — The Nonremovable, Windowed, Fiberglass Cast Boot is implemented before the beginning of CACIPLIQ20 treatment and is maintained during the treatment.
  CACIPLIQ20 is applied on the wound for 10 minutes every 3 to 4 days
  Arms: CACIPLIQ20 and Cast Boot
Device: Placebo and Nonremovable, Windowed, Fiberglass Cast Boot — The Nonremovable, Windowed, Fiberglass Cast Boot is implemented before the beginning of placebo treatment and is maintained during the treatment.
  Placebo is applied on the wound for 10 minutes every 3 to 4 days
  Arms: Placebo and Cast Boot

SUMMARY:
CACIPLIQ20 is a nanopolymer engineered to mimic glycosaminoglycans such as heparan sulfates. Glycosaminoglycans are implied 1) in the stabilization of the micro-environment of cells, known as extracellular matrix, by binding to structural proteins, and 2) in the cell communication by protecting growth factors. At the site of a lesion, glycosaminoglycans are degraded, thereby the extracellular matrix is disorganized and the tissue is destroyed. By replacing damaged glycosaminoglycans, CACIPLIQ20 provides a protective function and restores the matrix architecture and the cell communication, a process known as Matrix Therapy.

As for now, three non-controlled pilot studies have been carried out on small populations. They have shown a substantial enhancement of chronic wounds state after treatment with CACIPLIQ20. Therefore, the purpose of this new controlled study is to determine whether CACIPLIQ20 can shorten diabetic neuropathic plantar ulcers healing when the off-loading is mandatory.

The study's main hypothesis is that CACIPLIQ20 application on a non-healing diabetic plantar ulcer in an off-loading mandatory context would reinitiate the natural process of tissue regeneration and lead to total wound closure faster than following standard wound care.

DETAILED DESCRIPTION:
This study specifically targets diabetic patients presenting neuropathic plantar ulcers.

Diabetic patients have a 25% risk to develop foot ulcers during their life, and one diabetes-induced amputation is performed every 30 seconds in the world. Textbook-case of perforating foot ulcer (Malum Perforans Pedis) is caused by a mechanical impairment : only a thoroughly observed discharge may lead to good wound care and, ultimately, healing. Thus, this study proposes the utilization of an nonremovable windowed Fiberglass Cast Boot, a technique which has led to healing in 6 to 8 weeks for 95% of neuropathic foot ulcers treated that way.

As 80% of amputations are caused by non-healing ulcers, it appears obvious that enhancing foot wounds healing could reduce amputation rate and in that way fairly improve diabetic patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Perforating non-ischemic plantar ulcer with neuropathy in a diabetic patient
* Wound not healing for no less than 6 weeks, based on recruitment examination
* Wound surface spanning from 1 cm² to 10 cm²
* Foot off-loaded by a non-removable windowed, fiberglass cast boot
* Age of inclusion ≥ 18 years
* A contraceptive method must be used for women of childbearing age
* Realization of a preliminary physical examination

Exclusion Criteria:

* Wound not located on the foot, or ischemic, with edema, erythema, maceration or eczema
* Infection clinically approved (Fever, pus...)
* Osteitis
* Known hypersensitivity to heparin
* Treatment with Negative Pressure Wound Therapy within 30 days prior to enrollment
* Treatment ongoing or within 30 days prior to enrollment with growth factors or other biotechnology products
* Treatment ongoing or within 12 months prior to enrollment with hyperbaric oxygen therapy
* Patient with liver or kidney failure
* Patient with a known heavy condition that could require corticosteroid, anti-inflammatory or immunosuppressant treatments
* Patient already enrolled in a therapeutic clinical study focusing on an experimental molecule
* Pregnant or breastfeeding woman, or likely to be
* Non-affiliation to the French social security system
* Patient unable to attend to scheduled medical monitoring due to geographical, social or mental reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2014-01 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Kinetics of Evolution of wound size within 60 days | 60 days

SECONDARY OUTCOMES:
Evolution of remaining lesion rate | 8, 15, 30, 45 and 60 days
  Remaining lesion rate, defined as the ratio of lesion surface at the specified time to lesion surface before treatment, during time
Healing rate | 8, 15, 30, 45 and 60 days
  Healing rate, defined as the difference between two lesion rates at different times
Number of declared full wound healings | 8, 15, 30, 45 and 60 days
  Number of declared full wound healings during time, defined as non-oozing wound closure without any reopening after no less than 15 days, ascertained by the principal investigator and another member of his team
Number of wounds leading to amputation | 8, 15, 30, 45 and 60 days
  Number of wounds causing new amputations during time, as recorded after surgical measures sustained by patients
Pain experienced during time | Recruitment, 8, 15, 30, 45 and 60 days
  Pain experienced by patients, assessed with Numerical Rating Pain Scale (0 to 10) and amount of painkillers used

CONTACTS AND LOCATIONS:
Overall Officials: Georges Ha Van, MD, Principal Investigator — Pitié-Salpêtrière Hospital, Paris
Locations (1):
- Pitié-Salpêtrière Hospital, Paris, France